CLINICAL TRIAL: NCT06054880
Title: An Open-Label, Randomized, Multicenter Study to Evaluate the Safety, Efficacy, and Physician Satisfaction of Two Different Doses of Bludigo™ When Used as an Aid in the Determination of Ureteral Patency
Brief Title: Indigotindisulfonate Sodium Injection, USP as an Aid in the Determination of Ureteral Patency
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Prove pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: PVP-22IC04
Record Dates: First submitted 2023-08-30; First posted 2023-09-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ureter Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Saline (Placebo Comparator): 116 subjects treated with 5 ml of saline then crossover to treatment arm
  Interventions: Other: Saline injection 0.9%
- High Dose (Experimental): 58 subjects randomly treated with 5 mL of drug
  Interventions: Drug: Indigotindisulfonate sodium 0.8%; Other: Saline injection 0.9%
- Low Dose (Experimental): 58 subjects randomly treated with 2.5 mL of drug
  Interventions: Drug: Indigotindisulfonate sodium 0.8%; Other: Saline injection 0.9%

INTERVENTIONS:
Drug: Indigotindisulfonate sodium 0.8% — Experimental contrast dye that is commonly used as a visualization aid in pelvic and abdominal surgeries and for various diagnostic procedures in medical practice.
  Other Names: Bludigo
  Arms: High Dose; Low Dose
Other: Saline injection 0.9% — Placebo

SUMMARY:
This is a randomized, multicenter study to evaluate the efficacy and safety of two dose levels (2.5 mL and 5.0 mL) of Bludigo when used as an aid in the determination of ureteral patency.

DETAILED DESCRIPTION:
Subjects scheduled for a surgical procedure in which the patency of the ureter must be assessed by cystoscopy following the procedure, age 18 to 85 years inclusive, will be screened for participation. Screening will occur within 30 days before study drug administration (Day of Surgery). After signing the informed consent, review of inclusion and exclusion criteria will be performed, the collection of concomitant medications, medical history, physical examination, baseline laboratory testing, 12-lead ECG, and vital sign measurements will be completed during the screening visit.

On the day of surgery (Day 1) subjects will be evaluated for eligibility for randomization. Eligible subjects will be stratified by BMI (<30.0 kg/m2or ≥ 30.0 kg/m2) and randomized in a 1:1 ratio to receive a dose of either Bludigo™ high dose (5.0 mL) or Bludigo™ low dose (2.5 mL). Each randomized subject will serve as his/her own control (i.e., intra-patient controlled) by receiving a dose of normal saline prior to receiving the randomized Bludigo™ dose.

All treated subjects will have a follow-up visit 7 to 30 days (± 2 days) after the procedure. A final telephone follow-up call will occur on Day 30 (± 2 days) in subjects who have the follow-up visit before Day 28. Safety assessments will include monitoring of AEs during and post the procedure, clinical laboratory tests, 12-Lead ECG, and vital sign measurements.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between ≥ 18 and ≤ 85 years old
* Subjects who signed a written IRB approved, informed consent form
* Subjects scheduled for a surgical procedure in which the patency of the ureter must be assessed by cystoscopy following the procedure

Exclusion Criteria:

* Subjects with stage 4 or 5 Chronic Kidney Failure as evidenced by a GFR <30 mL/min (calculated using the MDRD formula and standardized by using individual's body surface area) or need for dialysis in the near future, or having only 1 kidney
* Subjects with known severe hypersensitivity reactions to Bludigo™ or other dyes, including contrast dyes
* Known history of drug or alcohol abuse within 6 months prior to the time of screening visit
* Subjects, as assessed by the Investigator, with conditions/concomitant diseases precluding their safe participation in this study (e.g. major systemic diseases)
* Unable to meet specific protocol requirements (e.g., scheduled visits) or subject is uncooperative or has a condition that could lead to non-compliance with the study procedures
* Subject is the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
* Subjects with life expectancy < 6 months
* Requirement for concomitant treatment that could bias primary evaluation.
* Subjects who are pregnant or breast-feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Paired sample difference (Bludigo™-Saline) in urine jet conspicuity score . | 10 minutes post study drug administration
  Visualization will be measured by a conspicuity scale designed to provide an objective tool applicable to the visualization of the urinary flow from the ureteral orifices when determining ureter patency. The conspicuity of the urine flow from the ureteral orifices is defined using the 5-point conspicuity score as follows:
  1. = No jet observed
  2. = Weak jet, little color contrast
  3. = Color contrast or significant jet flow
  4. = Strong jet flow with good color contrast
  5. = Strong jet flow with striking contrast in color
  Paired sample difference (Bludigo™-Saline) in conspicuity score (PSDCS). PSDCS will be calculated for each ureter (left or right) for each subject from each reviewer.
Responders to Bludigo | 10 Minutes post study drug administration
  Visualization will be measured by a conspicuity scale designed to provide an objective tool applicable to the visualization of the urinary flow from the ureteral orifices when determining ureter patency. The conspicuity of the urine flow from the ureteral orifices is defined using the 5-point conspicuity score as follows:
  1. = No jet observed
  2. = Weak jet, little color contrast
  3. = Color contrast or significant jet flow
  4. = Strong jet flow with good color contrast
  5. = Strong jet flow with striking contrast in color
  A subject is considered a responder to Bludigo™ if there is >=1 point improvement in the conspicuity score following the Bludigo™- treatment vs the saline treatment and the conspicuity score for the Bludigo™ treatment must be (3, 4, or 5). The responder criteria will be assessed separately for each ureter (left or right) from each reviewer.

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events. | 30 days post study drug administration
  Percentage of patients in each treatment group who experience an adverse event post treatment
Changes in clinical safety laboratory values | 30 days post study drug administration
  Proportion of subjects with clinically important changes in clinical safety laboratory tests after treatment
Changes in vital signs post treatment | 30 days post study drug administration
  Proportion of subjects with clinically important changes in vital signs after treatment
Changes in ECG post treatment | 30 days post study drug administration
  Proportion of subjects with clinically important changes in ECGs after treatment
Changes in blood pressure by dose group and BMI (kg/m^2) | 30 days post study drug administration
  Comparison of post treatment changes in blood pressure by dose group and BMI (kg/m^2)
Changes in heart rate by dose group and BMI (kg/m^2) | 30 days post study drug administration
  Comparison of post treatment changes in heart rate by dose group and BMI (kg/m^2)
Changes in pulse oximetry by dose group and BMI (kg/m^2) | 30 days post study drug administration
  Comparison of post treatment changes in pulse oximetry by dose group and BMI (kg/m^2)
Physician Satisfaction | 10 Minutes post study drug administration
  To determine physicians' overall satisfaction with the Bludigo™ treatment by assessing the proportion of surgeons who agree using the 5-point Physician Satisfaction Agreement Scale (PSAS) with the statement:
  "Compared to the saline treatment, my ability to assess ureter patency was improved after the addition of Bludigo™."
  1. = Strongly Agree
  2. = Agree
  3. = Neither Agree nor Disagree
  4. = Disagree
  5. = Strongly Disagree A surgeon's evaluation is considered satisfactory if the rating is either a 1 (strongly agree) or 2 (agree).
Time to visualization | 10 minutes post study drug administration
  To describe the time to visualization (TTV) of blue color in the ureteral jets flow following Bludigo™ treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Boytim, Ph.D., Study Director — Provepharm SAS
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No